CLINICAL TRIAL: NCT06786286
Title: A Phase 1, Open-label Study to Assess the Mass Balance, Metabolism, Excretion and Pharmacokinetics of a Single Subcutaneous Dose of [14C]-ITI-1284 in Healthy Male Subjects
Brief Title: A Mass Balance Study Following Subcutaneous Administration of [14C]-ITI-1284 to Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITI-1284-012
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]-ITI-1284 20 mg (Experimental)
  Interventions: Drug: [14C]-ITI-1284

INTERVENTIONS:
Drug: [14C]-ITI-1284 — [14C]-ITI-1284 20 mg oral solution (not more than 22 μCi), subcutaneous administration

SUMMARY:
ITI-1284-012 is an open-label, single-dose study to assess the mass balance recovery of radioactivity, and to evaluate the pharmacokinetics, safety and tolerability of ITI-1284 after a single subcutaneous dose of [14C]-ITI-1284 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between 30 and 55 years of age (inclusive);
* BMI between18.0 and 32.0 kg/m2, inclusive, at screening, and a minimum body weight of 50 kg at screening;
* Willing to be confined to the clinical research unit for the duration of the inpatient period of the study.

Exclusion Criteria:

* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposure, exceeding 5 mSev in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker shall participate in the study;
* Subjects who have been enrolled in a 14C-labeled product study in the 10 months prior to dosing with study drug on Day 1;
* Any clinical condition or procedure that may affect the absorption, distribution, biotransformation, or excretion of ITI-1284. Subjects with a history of appendectomy and/or abdominal wall hernia repair are eligible for study participation provided surgery was performed ≥1 year ago;
* Acute diarrhea or constipation in the 7 days before Day 1. If screening occurs > 7 days before Day 1, this criterion will be determined on Day 1;
* Clinically significant abnormal findings in vital sign assessments, supine SBP > 140 mmHg or < 90 mmHg, or supine DBP >90 mmHg or < 50 mmHg or supine pulse rate > 100 bpm or < 45 bpm at Screening;
* History of psychiatric condition that in the Investigator's opinion may be detrimental to participation in the study.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery of total radioactivity in urine and feces combined | Day 1 up to Day 29
  percentage of total radioactivity
Pharmacokinetics: AUC0-t for total radioactivity | Day 1 up to Day 29
  Area under the plasma drug concentration-time curve (AUC) from time zero to the last measurable concentration
Pharmacokinetics: AUC0-t for ITI-1284 | Day 1 to Day 8
  Area under the plasma drug concentration-time curve (AUC) from time zero to the last measurable concentration
Pharmacokinetics: Cmax for total radioactivity | Day 1 up to Day 29
  Maximum plasma concentration
Pharmacokinetics: Cmax for ITI-1284 | Day 1 to Day 8
  Maximum plasma concentration
Pharmacokinetics: Tmax for total radioactivity | Day 1 up to Day 29
  Time of maximum plasma concentration
Pharmacokinetics: Tmax for ITI-1284 | Day 1 to Day 8
  Time of maximum plasma concentration

SECONDARY OUTCOMES:
Percentage of subjects with treatment-emergent adverse events | Up to 30 days after the dose of study drug
Change from baseline in systolic and diastolic blood pressure | Day 14
Change from baseline in ECG QT interval | Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site 1, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No